CLINICAL TRIAL: NCT04116151
Title: Effectivenes and Safety of a Cream of Aloe Vera, Camomila and Tomillo (Alantel) for Profilaxis or Treatmment of Deratitis by Radiotheraphy in Patients With Breast Cancer
Brief Title: Effectiveness of a Cream for Treatment of Dermatitis in Patients Whith Breast Cancer
Acronym: Alantel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario Reina Sofia de Cordoba (Other Government)
Responsible Party: Principal Investigator, Luis A Perula, Clinical Professor, Hospital Universitario Reina Sofia de Cordoba
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Alantel
Record Dates: First submitted 2019-09-18; First posted 2019-10-04 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: DERMATITIS INDUCED BY RADIOTHERAPY IN PATIENTS WHITH BREAST CANCER
Keywords: BREAST CANCER; DERMATITIS
MeSH Terms: conditions — Breast Neoplasms; Dermatitis | interventions — Chamomile extract

STUDY DESIGN:
Intervention Model Description: Experimental, prospective, controlled clinical trial, with two parallel arms, double blind, multicenter study
Who Masked: Participant, Care Provider
Masking Description: Double blind: both the patient and the healthcare professional do not know if the cream to be tested or the placebo is applied
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Local administration of the Alantel (R) cream on the affected skin
  Interventions: Combination Product: Cosmetic cream (Alantel (R): aloe vera, chamomile and thime)
- Control group (Placebo Comparator): Local administration of the Placebo cream on the affected skin
  Interventions: Combination Product: Usual treatment

INTERVENTIONS:
Combination Product: Cosmetic cream (Alantel (R): aloe vera, chamomile and thime) — Application on the affected skin of the cream to be tested
  Arms: Intervention group
Combination Product: Usual treatment — Application on the affected skin of the emollient and moisturizing substance
  Arms: Control group

SUMMARY:
It is intended to evaluate the effect of a marketed cream (Alantel®) based on natural products at high concentrations for the preventive and curative treatment (early stages) of radiation-induced dermatitis in cancer patients. For this, an experimental, prospective, controlled clinical trial, with two parallel arms, double blind, multicentre, will be carried out in which doctors will recruit 78 patients aged 14 years or over in Primary Care consultations. more, diagnosed with cancer, and having received radiotherapeutic cancer treatment, being randomly assigned to the experimental group (cosmetic cream) or the control group (emollient and moisturizing cream). The main variable will be the incidence rate of mild post-translational dermatitis and its improvement or cure once it has been established.

ELIGIBILITY:
Inclusion Criteria:

* Patients 14 years of age or older
* Diagnosed with cancer and who are or have recently received radiotherapy treatment.
* We will include patients without dermatitis or with acute dermal posttradiotherapy lesions, in grades 1 and 2.

Exclusion Criteria:

* Patients with dermal lesions in grade greater than 2.
* Skin cancer invasion or distant tumor metastasis.
* Concurrent chemotherapy with RT, severe / extensive burns, moisture, erosion or suppuration in the skin, history of connective tissue disorders, severe mental disorder (dementia, drug addiction, etc.).
* History of hypersensitivity reaction to any of the ingredients of the studio cream.
* Participants involved in other clinical trials within that month.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2022-07-19 (Actual); Primary Completion 2023-05-30 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Incidence of radiation-induced dermatitis | three weeks
Analog visual scale | three weeks
  Analog visual scale from 0 to 10 points to assess the symptomatology perceived by the patient (pain, stinging, ..)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Cordoba, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jimenez-Garcia C, Perula-de Torres LA, Villegas-Becerril E, Munoz-Gavilan JJ, Espinosa-Calvo M, Montes-Redondo G, Romero-Rodriguez E; Alantel Trial Collaborative Group. Efficacy of an aloe vera, chamomile, and thyme cosmetic cream for the prophylaxis and treatment of mild dermatitis induced by radiation therapy in breast cancer patients: a controlled clinical trial (Alantel Trials). Trials. 2024 Jan 25;25(1):84. doi: 10.1186/s13063-024-07901-8. PMID 38273379